CLINICAL TRIAL: NCT07377435
Title: Phase I Study of Vaccination With DC/MM Fusion Cells in Combination With BCMA Directed CAR-T Cell Therapy in Relapsed/Refractory Multiple Myeloma
Brief Title: DC/MM Fusion Vaccine With BCMA CAR-T in R/R MM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Avigan (Other)
Collaborators: The V Foundation (Other)
Responsible Party: Sponsor-Investigator, David Avigan, Sponsor-Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-799
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma; Relapse Multiple Myeloma
Keywords: Multiple Myeloma; Refractory Multiple Myeloma; Relapsed Multiple Myeloma; MM
MeSH Terms: conditions — Multiple Myeloma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DC/MM Fusion Vaccine: (Experimental): 25 participants will be enrolled and will complete the following:
  * Baseline visit
  * Leukapheresis for dendritic and tumor cell collection
  * Standard of care BCMA CAR-T cell therapy
  * Cycles 1 through 2 (28 day cycle):
    --Day 1: predetermined dose of DC/MM Fusion Vaccine 1x daily and predetermined dose of GM-CSF 1x daily
  * Follow up every 3 months starting at month 12 to year 5
  Interventions: Biological: DC/MM Fusion Vaccine; Drug: GM-CSF

INTERVENTIONS:
Biological: DC/MM Fusion Vaccine — Dendritic Cell and tumor fusion vaccine, via subcutaneous injection (under the skin), per protocol.
  Other Names: Dendritic Cell and Tumor Fusion Vaccine
Drug: GM-CSF — Granulocyte-Macrophage Colony-Stimulating Factor, via subcutaneous injection, per standard of care.
  Other Names: Granulocyte-Macrophage Colony-Stimulating Factor

SUMMARY:
This study is to evaluate the safety and effectiveness of dendritic cell DC/MM fusion vaccine in combination with standard of care B-cell maturation antigen (BCMA) CAR-T cell therapy in participants with relapsed/refractory multiple myeloma.

The names of the study drugs involved in this study are:

* DC/MM fusion vaccine (a type of personalized cancer vaccine)
* Granulocyte-macrophage colony-stimulating factor (GM-CSF) (a type of growth factor or hormone)

DETAILED DESCRIPTION:
This Phase I study is to evaluate the safety and effectiveness of dendritic cell DC/MM fusion vaccine in combination with standard of care B-cell maturation antigen (BCMA) CAR-T cell therapy in participants with relapsed/refractory multiple myeloma. The DC/MM fusion vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells.

The U.S. Food and Drug Administration (FDA) has not approved DC/MM fusion vaccine as a treatment for relapsed or refractory multiple myeloma.

The FDA has approved GM-CSF as a treatment for relapsed or refractory multiple myeloma.

The research study procedures include screening for eligibility, in-clinic visits, collection of dendritic and tumor cells in a process called leukapheresis, blood tests, urine tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans, X-rays, electrocardiograms (ECGs), bone marrow biopsies and aspirations.

It is expected about 25 people will take part in this research study.

The V Foundation for Cancer Research is providing funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be eligible to receive standard of care CAR T-cell therapy for relapsed or refractory multiple myeloma
* Patients must be ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients must have 20% or more plasma cells in the bone marrow core or aspirate differential within 30 days prior to enrollment.
* Patients must have adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 x institutional upper limit of normal
  * AST ≤ 3 x institutional upper limit of normal
  * ALT ≤ 3 x institutional upper limit of normal
  * Creatinine clearance ≥ 40 mL/min for participants with creatinine levels above institutional normal
* The effects of DC/MM fusion vaccine on the developing human fetus are unknown. For this reason, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier methods of birth control or abstinence) prior to study enrollment and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of treatment.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients receiving other investigational drugs
* Patients with Plasma Cell Leukemia

  * Patients who have known active uncontrolled infections with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV)
  * Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias. Prior to study entry, any ECG abnormality at screening will be documented by the investigator as not medically relevant.
* Female patients who are pregnant (positive β-HCG) or breastfeeding.
* Prior organ transplant requiring immunosuppressive therapy.
* Uncontrolled intercurrent illness including, but not limited to: active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of intolerance to CAR-T related drugs or GM-CSF.

Inclusion Criteria Prior to Vaccination with DC/MM Fusions:

* Resolution of all CAR T- related grade 3-4 toxicities
* Successful production of at least 2 vaccines with a minimum of 1 x 106 fusion cells
* Absence of disease progression following CAR T-cell therapy
* ECOG performance status ≤ 2
* Patients must have adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 x institutional upper limit of normal
  * AST ≤ 3 x institutional upper limit of normal
  * ALT ≤ 3 x institutional upper limit of normal
  * Creatinine within normal limits or Creatinine clearance ≥ 40 mL/min for participants with creatinine levels above institutional normal
  * ANC >1000 in the absence of growth factor support in the prior 7 days
  * Platelet count >50K without the need for transfusion in the prior 7 days
  * No myeloma-directed therapy following administration of CAR T-cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Limiting Toxicity (TLT) Rate | Assessed 28 days post-vaccination.
  TLT rate, defined as the proportion of participants who experience treatment-limiting toxicity (TLT) as detailed in Protocol Section 6.1.
Vaccine/Granulocyte-Macrophage Colony-Stimulating Factor(GM-CSF)-Related Adverse Event (AE) Rate | Assessed during the vaccination period of 8 weeks and then up to 1 year post-vaccination.
  Vaccine/GM-CSF-related AE rate is defined as the proportion of participants who experience any grade AE deemed by investigators as possibly, probably, or definitely related to vaccine or GM-CSF based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Grade 3 or 4 Cytokine Release Syndrome (CRS) Rate | Assessed during the vaccination period of 8 weeks and then up to 1 year post-vaccination.
  Grade 3 or 4 CRS rate is defined as the proportion of participants who experience grade 3 or 4 CRS based on the American Society of Transplantation and Cellular Therapy (ASTCT) consensus guidelines.
Grade 3 or 4 Immune-effector Cell-associated Neurotoxicity (ICANS) Rate | Assessed during the vaccination period of 8 weeks and then up to 1 year post-vaccination.
  Grade 3 or 4 ICANS rate is defined as the proportion of participants who experience grade 3 or 4 ICANS based on the American Society of Transplantation and Cellular Therapy (ASTCT) consensus guidelines.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | 12 months
  CR rate is defined as the proportion of participants who experience CR or stringent CR per International Myeloma Working Group (IMWG) Uniform Response Criteria.
Measurable Residual Disease (MRD) Negative Rate | 12 months
  Measurable Residual Disease (MRD) Negative Rate is defined as the proportion of patients who achieve MRD negativity, as assessed by clonoSEQ. Participants who receive at least 1 dose of the vaccine will be included in the analysis.
Progression-Free Survival (PFS) at 12 months | 12 months post-CAR-T cell therapy
  PFS based on Kaplan-Meier method is defined as the time from registration to the earlier of progression per International Myeloma Working Group (IMWG) Uniform Response Criteria or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu